CLINICAL TRIAL: NCT07075341
Title: Healthy Living BEYOND Weight Study
Status: Recruiting | Type: Observational
Sponsor: American Heart Association (Other)
Collaborators: Evidation Health (Industry); Duke Clinical Research Institute (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00086052
Record Dates: First submitted 2025-06-03; First posted 2025-07-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Overweight or Obesity
Keywords: overweight; obesity; weight management; BMI; cardiovascular disease; Cardiovascular-Kidney Metabolic; CVD; CKM; GLP-1 RA; glucagon-like peptide-1; GLP-1; GLP-1 receptor agonists; bariatric
MeSH Terms: conditions — Overweight; Obesity; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Direct-to-Participant Group: Observational
  Interventions: Other: None - Observational study

INTERVENTIONS:
Other: None - Observational study — None - Observational study

SUMMARY:
The Healthy Living BEYOND Weight Study is an observational research study of participants living with overweight and obesity. The principal objectives for this project will be to answer fundamental unanswered questions regarding patient experiences and outcomes related to overweight and obesity, and to assess the real-world effectiveness of different weight management strategies, within contemporary and diverse populations. To accomplish this, the Study Team for this project will leverage their expertise in the science of obesity and cardiometabolic health; epidemiology, cohort and registry studies; implementation science; cardiovascular prevention and management; and disparities and community-based research to lead the development of an innovative cohort of people living with overweight or obesity with two key components:

1. patient-report data elements, obtained through surveys;
2. linkage to EHR records providing data regarding clinical encounters.

The cohort will be inclusive, comprehensive, and constructed with scientific rigor as well as high internal and external validity. An overall objective is for the Healthy Living BEYOND Weight Study is to serve as an enduring resource for researchers studying the health consequences of obesity and evaluating the impact of weight management strategies.

DETAILED DESCRIPTION:
Obesity and overweight are presently the leading clinical and public health challenge in the United States. Nationally representative data demonstrates a historically high domestic prevalence of obesity, with a disproportionately high burden in vulnerable populations. There are myriad clinical consequences of obesity, with the most significant adverse impact being premature mortality due to an excess burden of cardiovascular disease. The cardiovascular consequences of overweight and obesity are mediated through cardiovascular-kidney-metabolic syndrome, involving multisystem dysfunction and progressive vascular pathology. While the public health urgency of overweight and obesity is well established, the landscape of obesity management has been revolutionized in recent years by the emergence of increasingly effective and safe obesity pharmacotherapies, in addition to refined approaches to lifestyle modification and bariatric surgery. Clinical trials and observational studies have demonstrated the efficacy of these obesity therapies for inducing weight loss, improving Cardiovascular-Kidney Metabolic (CKM) risk factor profiles and decreasing rates of adverse kidney and cardiovascular events. However, many substantial questions remain regarding the real world and long-term utilization and impact of these therapies, as well as the broader lived experience of individuals living with overweight and obesity. Utilizing direct engagement with participants and the examination of health records, the Healthy Living BEYOND Weight Study is poised to provide important new insights about the health, well-being and approaches to care for persons living with overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* BMI at the time of enrollment of 25 kg/m2 or greater or other elevated adiposity measures (e.g., waist circumference of greater than 102cm (40 in) in men or 88cm (35 in) in women) OR adults with a BMI less than 25 due to previous or current weight management treatment (lifestyle, pharmacological or surgical).

Exclusion Criteria:

* Incarcerated at the time of enrollment
* Self-reported pregnancy at the time of enrollment. However, individuals who become pregnant after enrollment will be welcomed to continue to participate, given that the critical life period of pregnancy often has a significant impact on subsequent weight trajectories.
* Terminal illness or end-stage disease with a life expectancy of less than 6-months
* Employed by the American Heart Association or working on the Healthy Living BEYOND Weight Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals currently residing in the United States
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2060-12 (Estimated); Study Completion 2060-12 (Estimated)

PRIMARY OUTCOMES:
Answer fundamental unanswered questions regarding patient experiences and outcomes related to overweight and obesity. | From enrollment to at least 10 years post enrollment, continuous follow up
Evaluate the real-world effectiveness of different weight management strategies, within contemporary and diverse patient populations. | From enrollment to at least 10 years post enrollment, continuous follow up
Create a community of volunteers interested in advancing research on the conditions of overweight/obesity and related weight management strategies. | From enrollment to at least 10 years post enrollment
To provide an enduring resource of value to individuals living with overweight and obesity. | From enrollment to at least 10 years post enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- American Heart Association, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from surveys will be combined with data from the EHR. Data that are stored in the integrated study database will use unique participant identification numbers, with data otherwise de-identified. We will utilize multiple data quality control processes to ensure the accuracy and reliability of study data. The integrated database will be maintained by the AHA or another service provider that is approved in advance by the IRB. Data collected as part of the Healthy Living BEYOND Weight Study will be used for research purposes only and will not be used for diagnosis or disease management.
Supporting Information: Study Protocol, ICF
Time Frame: July 2026 - ending 5 years after study close
Access Criteria: Study participant de-identified data will be accessible by the AHA and organizations doing work on their behalf such as qualified researchers, academic institutions, patient-advocacy groups, pharmaceutical, medical device companies, Evidation Health, Inc., and more. Study participant de-identified data may be used for the following:
  * Determination of clinical Study eligibility and subsequent screening, recruitment and enrollment. If a participant chooses to join a clinical Study for which they are eligible, they may be asked to sign an additional Study-specific consent form.
  * Use for research across a variety of disciplines and for use in scientific publications, interventional and/or product development.
  Data will be stored in a HIPAA-compliant, secure electronic platform with access limited to authorized study personnel and authorized researchers with executed data use agreements.
URL: https://www.heart.org/gobeyond

REFERENCES:
- See also: Related Info — https://www.heart.org/en/healthy-living/healthy-living-beyond-weight-study